CLINICAL TRIAL: NCT00066742
Title: A Phase II Study of Tirapazamine (NSC-130181)/Cisplatin/Etoposide and Concurrent Thoracic Radiotherapy for Limited Stage Small Cell Lung Cancer
Brief Title: Tirapazamine Combined With Chemo and RT in Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03042; NCI-2012-03042 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA032102 (NIH); S0222 (Other: SWOG); S0222 (Other: CTEP)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2012-07-19 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2012-12

CONDITIONS: Limited Stage Small Cell Lung Cancer
MeSH Terms: interventions — Tirapazamine; Cisplatin; Etoposide; Radiotherapy; Radiation

ARMS (1):
- Treatment (tirapazamine, cisplatin, etoposide) (Experimental): CHEMORADIOTHERAPY: Patients receive tirapazamine IV over 1 hour on days 1, 8, 10, 12, 29, 36, 38, and 40; cisplatin IV over 1 hour on days 1, 8, 29, and 36; and etoposide IV over 1 hour on days 1-5 and 29-33. Beginning on day 1 of chemotherapy, patients undergo thoracic radiotherapy once daily 5 days a week for 7 weeks.
  CONSOLIDATION CHEMOTHERAPY: Within 28 days after completion of radiotherapy, patients with stable or responding disease receive cisplatin IV over 1 hour on days 1 and 22 and etoposide IV over 1 hour on days 1-3 and 22-24.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tirapazamine; Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tirapazamine — Given IV
  Other Names: SR 4233; Tirazone; WIN 59075
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving tirapazamine together with cisplatin, etoposide, and radiation therapy works in treating patients with limited-stage small cell lung cancer. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Tirapazamine may make the tumor cells more sensitive to chemotherapy and radiation therapy. Combining chemotherapy and radiation therapy with tirapazamine may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess overall survival in patients with limited stage small cell lung cancer (SCLC) treated with induction tirapazamine combined with cisplatin, etoposide and high dose thoracic radiotherapy followed by consolidative cisplatin and etoposide.

II. To assess time to treatment failure calculated from initiation of step 1, response (confirmed plus unconfirmed, complete plus partial during induction in the subset of patients with measurable disease) and toxicity in this patient population treated with this regimen.

III. To investigate in an exploratory manner the association of baseline PAI-1, VEGF, OPN and NDRG1 plasma markers with patient response and survival.

OUTLINE: This is a multicenter study.

CHEMORADIOTHERAPY: Patients receive tirapazamine IV over 1 hour on days 1, 8, 10, 12, 29, 36, 38, and 40; cisplatin IV over 1 hour on days 1, 8, 29, and 36; and etoposide IV over 1 hour on days 1-5 and 29-33. Beginning on day 1 of chemotherapy, patients undergo thoracic radiotherapy once daily 5 days a week for 7 weeks.

CONSOLIDATION CHEMOTHERAPY: Within 28 days after completion of radiotherapy, patients with stable or responding disease receive cisplatin IV over 1 hour on days 1 and 22 and etoposide IV over 1 hour on days 1-3 and 22-24.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2-3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 30-85 patients will be accrued for this study within 17 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of limited small cell lung cancer; diagnosis on the basis of sputum cytology is acceptable if confirmation by an independent pathologic review at the institution is documented
* Patients must have measurable OR non-measurable disease documented by CT, MRI or X-ray; any scan abnormalities, which may otherwise represent metastatic disease, should be confirmed benign by appropriate tests and documented on the baseline tumor assessment form (form #848); if an abnormality is present at baseline, it is assumed to be disease involvement unless proven otherwise; disease must be assessed within 28 days prior to registration for measurable disease and 42 days prior to registration for non-measurable disease; NOTE: The use of PET scans for tumor imaging is not allowed
* Patients with any brain metastases are ineligible; all patients must have a pretreatment CT or MRI scan of the brain to evaluate CNS disease within 42 days prior to registration
* Patients with malignant pericardial effusions OR malignant pleural effusions are ineligible; these are defined as either cytologically positive effusions OR exudative effusions not attributable to other etiologies; patients with effusions too small to tap are eligible
* Patients must have a measured or calculated creatinine clearance >= 50 cc/min obtained within 28 days prior to registration; serum creatinine is only necessary if calculated CrCl is used; if calculated CrCl is used, serum creatinine must be < 1.5 mg/dl
* ANC >= 1,500/ul obtained within 28 days prior to registration
* Platelet count >= 100,000/ul obtained within 28 days prior to registration
* Serum bilirubin =< 1.5 x the institutional upper limit of normal within 28 days prior to registration
* SGOT or SGPT =< 2 x the institutional upper limit of normal within 28 days prior to registration
* All patients must have a Zubrod performance status of 0-1
* Patients must not have received previous chemotherapy or biologic therapy for small cell lung cancer; patients must not have received prior thoracic or neck radiation for any reason
* At least two weeks must have elapsed since surgery (thoracic or other major surgeries) and patients must have recovered from all associated toxicities; measurable or non-measurable disease must be present outside the area of surgical resection
* Patients with significant clinical hearing loss must be willing to accept the potential for worsening of symptoms
* Patients must not have >= grade 1 symptomatic neuropathy-sensory (NCI Common Terminology Criteria for Adverse Events version 3.0)
* Patients must have a pre-registration FEV1 and DLCO obtained within 28 days prior to registration
* Institutions must have received IRB approval of S9925 (the Lung Cancer Specimen Repository); patients must be offered participation in S9925; with the patient's consent, plasma, serum and tissue will be submitted for testing via S9925; patients must be registered separately to S9925 to receive credit for specimen submission
* The radiation oncology facility must be willing to deliver 3D conformal radiation; if the radiation therapy is to be done at a different institution, then the institution name and ID must be provided; the radiation therapy facility must be SWOG-approved; NOTE: The radiation oncology facility must have successfully completed the benchmark material from the Quality Assurance Review Center (QARC) or be willing to complete the benchmark material prior to submission of the final radiation forms due within 30 days of completing radiation therapy
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for at least 5 years
* If day 28 or 42 falls on a weekend of holiday, the limit may be extended to the next working day; in calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday four weeks later would be considered day 28; this allows for efficient patient scheduling without exceeding the guidelines
* Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including fetal death from the chemotherapeutic agents; women of reproductive potential must have agreed to use an effective contraceptive method
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the times of patient registration, the treating institution's name and ID number must be provided to the Data Operation Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the database

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group (SWOG) Research Base, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 9/2003 and 7/2006, 72 of planned 85 limited smal-cell lung cancer patients were enrolled by SWOG institutions. The study was closed early due to a report of excess toxicity for Tirapazamine in a head and neck cancer trial elsewhere.
Groups:
- Evaluable Patients: Only eligible patients who received the study intervention were included in the analysis.
Period: Induction Chemoradiotherapy
Arm/Group | Evaluable Patients
Started | 72
Eligible | 69
Began Protocol Treatment | 68
Completed | 43
Not Completed | 29
Not completed — Did not receive any protocol treatment | 1
Not completed — Adverse Event | 21
Not completed — Withdrawal by Subject | 2
Not completed — not protocol specified | 2
Not completed — Ineligible | 3
Period: Consolidation Chemotherapy
Arm/Group | Evaluable Patients
Started | 42
Eligible | 40
Completed | 39
Not Completed | 3
Not completed — not protocol specified | 1
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 68
Age, Continuous [Median (Full Range); unit: years] | 63 [39 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 63
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from date of enrollment until the date of death due to any cause. Patients last known to be alive were censored at the date of last conatct. Patients were followed for a maximum of 3 years from the date of enrollment.
Time Frame: Weekly during protocol treatment, then every 3 months for first year, then every 6 months for up to 3 years after enrollment.
Population: Only eligible patients who received protocol treatment were included in the analsysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 68
months | 21 [17 to 32]

2. Secondary Outcome: Response Rate (Confirmed and Unconfirmed Complete and Partial Responses Per RECIST) in the Subset of Patients With Measurable Disease at Baseline.
Description: A complete response (CR) was defined as a complete disappearance of all disease with no new lesions. A partial response (PR) was defined as at least a 30% decrease under baseline of the sum of longest diameters of all target measurable lesions with no unequivocal progression of non-measurable disease and no new lesions. Both CR and PR had to be confirmed by a second determination at least 4 weeks apart. All disease had to be assessed using same method as baseline. Only patients with measurable disease at baseline were included in this analysis.
Time Frame: After completeion of concurrent chemotherapy+radiation (Week 8); then after completion of consolidation chemotherapy (Week15); once off treatment, every 3 months until disease progression for a maximum of 3 years after enrollment.
Population: Only eligible patients who received protocol treatment were included in the analysis.
Measure: Number; unit: participants
Groups:
- Evaluable Patients With Measurable Disease: Only eligible patients who received protocol treatment and who had measurable lesions (per RECIST) at baseline were included in this analysis.
Arm/Group | Evaluable Patients With Measurable Disease
Number analyzed (Participants) | 63
participants
  Complete Response | 0 [49% to 74%]
  Unconfirmed Complete Response | 7
  Partial Response | 2
  Unconfirmed Partial Response | 30
  No response | 24

3. Secondary Outcome: Progression-Free Survival
Description: Progression was defined as a >= 20% increase in the sum of longest diameters of measurable lesions over the smallest sum observed or unequivocal progression of non-measurable disease or the appearance of any new lesion/site. Symptomatic deterioration was defined as a global deterioration of health status requiring discontinuation of treatment. Progression-free survival was defined as the time from the date of enrollment until the date of progression, symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free were censored at last contact date.
Time Frame: At end of concurrent chemoradiotherapy (Week 8), then at end of consolidation chemotherapy (Week 15). After off treatment, every 3 months for the first 2 years then every 6 months for up to 3 years after enrollment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 68
months | 11 [10 to 13]

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events weekly during concurrent radiotherapy, and every 3 weeks during consolidation chemotherapy.
Description: This study utilized the CTCAE (NCI Common Toxicity Criteria for Adverse Events) version 3.0
Arm/Group | Tirapazamine + Cisplatin + Etoposide + Concurrent Radiotherapy | Consolidation Cisplatin + Etoposide
Serious Adverse Events (participants affected / at risk) | 24/68 | 5/39
Other Adverse Events (participants affected / at risk) | 67/68 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirapazamine + Cisplatin + Etoposide + Concurrent Radiotherapy (N=68) | Consolidation Cisplatin + Etoposide (N=39)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 | 0
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 | 0
Esophagitis (Gastrointestinal disorders) | 7 | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI - Esophagus (Gastrointestinal disorders) | 0 | 1
Mucositis/stomatitis (clinical exam) - Esophagus (Gastrointestinal disorders) | 1 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 | 0
Pain - Esophagus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 0
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 1 | 0
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 0 | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Catheter-rela (Infections and infestations) | 1 | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (pneumon (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Soft tissue NOS (Infections and infestations) | 1 | 0
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 | 0
Leukocytes (total WBC) (Investigations) | 6 | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7 | 1
Platelets (Investigations) | 4 | 2
Weight loss (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 13 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 | 0
Death not associated with CTCAE term - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (fainting) (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tirapazamine + Cisplatin + Etoposide + Concurrent Radiotherapy (N=68) | Consolidation Cisplatin + Etoposide (N=39)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 4
Hemoglobin (Blood and lymphatic system disorders) | 49 | 32
Tinnitus (Ear and labyrinth disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 32 | 8
Diarrhea (Gastrointestinal disorders) | 22 | 6
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 32 | 13
Esophagitis (Gastrointestinal disorders) | 32 | 12
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 5 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 2
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5 | 3
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 13 | 6
Nausea (Gastrointestinal disorders) | 49 | 18
Pain - Abdomen NOS (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 30 | 11
Fatigue (asthenia, lethargy, malaise) (General disorders) | 54 | 30
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 8 | 4
Rigors/chills (General disorders) | 6 | 3
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (pneumon (Infections and infestations) | 0 | 2
Rash: dermatitis associated with radiation - Radiation (Injury, poisoning and procedural complications) | 15 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 10 | 2
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 5 | 0
Alkaline phosphatase (Investigations) | 5 | 2
Bilirubin (hyperbilirubinemia) (Investigations) | 4 | 0
Creatinine (Investigations) | 7 | 4
Leukocytes (total WBC) (Investigations) | 52 | 30
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 48 | 30
Platelets (Investigations) | 41 | 24
Weight loss (Investigations) | 26 | 13
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 9 | 2
Anorexia (Metabolism and nutrition disorders) | 10 | 6
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 19 | 7
Dehydration (Metabolism and nutrition disorders) | 21 | 9
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 11 | 6
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 19 | 9
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 7 | 7
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8 | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 6 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 32 | 8
Neuropathy: sensory (Nervous system disorders) | 8 | 6
Taste alteration (dysgeusia) (Nervous system disorders) | 19 | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 45 | 26
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 | 0
Hypotension (Vascular disorders) | 14 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less